CLINICAL TRIAL: NCT00260533
Title: Double Blind Placebo Controlled Parallel Group Comparison of Atomoxetine (Strattera) for Generalized Social Anxiety Disorder (GSAD)
Brief Title: Efficacy and Tolerability of Atomoxetine (Strattera) in Adult Patients With Generalized Social Anxiety Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Murray B. Stein, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 040100
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Generalized Social Phobia
MeSH Terms: interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atomoxetine
  Interventions: Drug: atomoxetine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atomoxetine — Flexible dose, up to 50 mg per day
  Other Names: Strattera
  Arms: 1
Drug: placebo — placebo (matching to atomoxetine)
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness and tolerability of atomoxetine (Strattera) in adult patients with generalized social anxiety disorder (an anxiety disorder characterized by a fear of interpersonal interactions).

DETAILED DESCRIPTION:
Controlled studies show that approximately 50% of patients with generalized social anxiety disorder(GSAD)will respond to treatment with available pharmacotherapeutic agents such as SSRI's. This still leaves 50% that respond partially or not at all. Those who do respond, often experience adverse events (e.g., sexual dysfunction), which leads them to discontinue treatment. Thus, there is a strong rational for identifying alternatives to SSRI's that are effective with fewer side effects (or with a different side-effect profile, that features less sexual dysfunction)for the treatment of GSAD. Available data demonstrate that sustained-release venlafaxine, a dual reuptake inhibitor, is also effective for GSAD.(Stein et al., 2005). It is unclear from these studies whether serotonin reuptake is integral to efficacy for social anxiety disorder, or whether norepinephrine reuptake will convey similar efficacy. Atomoxetine (Strattera)an inhibitor of the presynaptic norepinephrine transporter, is an ideal candidate to address both these issues.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women, ages 18-65, in good general health
* Meet DSM-IV criteria for Social Anxiety Disorder

Exclusion Criteria:

* Pregnant or breastfeeding
* Narrow angle glaucoma
* Any uncontrolled medical condition or any medical condition which would represent a contraindication to atomoxetine (Strattera) pharmacotherapy (e.g., hepatic insufficiency, untreated hypertension, untreated cardiovascular or cerebrovascular disease)
* Any concomitant non-psychotropic medications that the physician determines are a contraindication to atomoxetine (Strattera) pharmacotherapy (e.g., Albuterol, various pressor agents)
* Bipolar disorder, or any psychotic or organic mental disorder or dementia
* Current substance abuse or dependency
* Current active suicidal ideation
* Current use of herbal psychoactive treatments such as St. John's Wort
* Concurrent psychotropic medication is not permitted for 2 weeks prior to randomization (4 weeks in the case of fluoxetine) or at any point thereafter.
* Receipt of formal psychotherapy concurrently
* Inability, in the investigator's opinion, to comply with study procedures or assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, M.D., Principal Investigator — University of California, San Diego

REFERENCES:
- [Result] Ravindran LN, Kim DS, Letamendi AM, Stein MB. A randomized controlled trial of atomoxetine in generalized social anxiety disorder. J Clin Psychopharmacol. 2009 Dec;29(6):561-4. doi: 10.1097/JCP.0b013e3181bf6303. PMID 19910721
- See also: UCSD Anxiety Disorders Research Program — http://www.veryshy.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient recruitment.
Groups:
- Atomoxetine: Atomoxetine 40-100 mg per day
- Placebo: Placebo (matched capsules to atomoxetine)
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 14 | 13
Completed | 11 | 10
Not Completed | 3 | 3
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine: Atomoxetine
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression (Change Version, Also Known as Improvement Version)
Description: This is a commonly used, clinician-rated measure of clinical improvement.
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
  For purposes of analysis, subjects rated as "(1) Very Much Improved" or "(2) Much Improved" were considered "responders".
Time Frame: 10 weeks (end of study)
Measure: Number; unit: participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 13
participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

LIMITATIONS AND CAVEATS:
Small study, with possibility of Type II error. Nonetheless, response rates in both arms were very low, making it unlikely that the failure to see a response to atomoxetine was due to low power compared to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No